CLINICAL TRIAL: NCT06913114
Title: Exploring the Relationship Between Hip Extensor Strength and Gait Speed in Diplegic Cerebral Palsy: A Feasibility Pilot Study
Brief Title: Relationship Between Hip Extensor Strength and Gait Speed in Diplegic Cerebral Palsy
Status: Active, not recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Abd Elaziz Anter, Lecturer, Cairo University
Other Study IDs: P.T.REC/012/005620
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Diplegic Spastic Cerebral Palsy
MeSH Terms: conditions — Cerebral palsy, spastic, diplegic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- study group
  Interventions: Diagnostic Test: Lafayette

INTERVENTIONS:
Diagnostic Test: Lafayette — The Lafayette handheld dynamometer data correlates with the measurements taken using the 10-Meter Walk Test (10MWT) or not.
Diagnostic Test: Lafayette — Lafayette handheld dynamometer.

SUMMARY:
The hip extensors are essential for upright posture and forward propulsion during gait. Children with diplegic CP often demonstrate reduced muscle strength, which impacts their gait speed and overall mobility. Understanding the relationship between hip extensor strength and gait speed could provide a basis for targeted interventions. This feasibility study will establish whether the handheld dynamometer can reliably measure hip extensor strength and if this strength correlates with gait speed in children with diplegic CP.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosed with diplegic CP

  * Ages 6 - 8 years
  * GMFCS Levels I-II (indicating they are ambulatory)
  * Able to follow instructions and participate in strength and gait assessments

Exclusion Criteria:

* • Severe cognitive or behavioral impairments affecting participation

  * Musculoskeletal conditions or recent orthopedic surgery that could interfere with hip function
  * Use of assistive devices for ambulation

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with diplegic CP who can walk
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Hip Extensor Strength | 4 months
  Hip extensor strength measured using a Lafayette handheld dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Faculty of Physical Therapy, Cairo, Egypt